CLINICAL TRIAL: NCT05920980
Title: Effect of Perioperative Continuous Intravenous Infusion of Lidocaine on Postoperative Pain in Elderly Patients Undergoing Colorectal Cancer Surgery: a Prospective, Randomized Controlled Trial
Brief Title: Effect of Lidocaine on Postoperative Pain in Elderlypatients Undergoing Colorectal Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chunling Jiang, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020HX1180
Record Dates: First submitted 2023-06-02; First posted 2023-06-27 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: Patients were randomized in a 1:1 lidocaine group, placebo control group using a computer-generated random number table. After the randomization scheme is written, use the opaque envelope, hide each group envelope into an opaque envelope, the envelope outside the code, is sealed to the researcher, when the study, if the inclusion criteria, then open the corresponding numbered envelope, and intervene according to the group scheme in the envelope.
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding of research personnel and patients will be maintained throughout the observation period. On the day of surgery, nurses who did not participate in the perioperative management will assign the standard configuration of the trial drugs, including intraoperative medication and the configuration of the postoperative analgesic pump, to the researchers before the induction of anesthesia. Throughout the study, the patients and researchers should not be unblinded until the statistical analysis of the study data is completed.
  During the operation, an independent anesthesiologist will be responsible for the blood draw, and the postoperative blood samples will be collected together with the routine blood examination specimens. The investigators remained blinded throughout the observation period until the anesthesiologist or assessors observe significant adverse events of local general anesthesia toxicity.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine group (Experimental): Patients in the lidocaine groups, lidocaine 1.5mg/kg/h was continuously infused (using ideal body weight) during the whole procedure, postoperative analgesia pump with lidocaine (lidocaine 50mg/kg, sufentanil 2ug/kg, glassetron 12mg), diluted to 200ml with saline until 72h after surgery. Blood samples will be collected from some patients in the lidocaine group for the measurement of lidocaine plasma concentration.
  Interventions: Drug: lidocaine
- Placebo group (Placebo Comparator): In the placebo group, the same volume of normal saline will be administered during anesthesia. The postoperative PCIA device will contain sufentanil 2 μg/kg, granisetron 12 mg diluted to 200 mL in 0.9% normal saline solution with a total volume of 200 mL.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: lidocaine — Patients in the lidocaine groups, lidocaine 1.5mg/kg/h was continuously infused (using ideal body weight) during the whole procedure, postoperative analgesia pump with lidocaine (lidocaine 50mg/kg, sufentanil 2ug/kg, glassetron 12mg), diluted to 200ml with saline until 72h after surgery. Blood samples will be collected from some patients in the lidocaine group for the measurement of lidocaine plasma concentration.
  Arms: Lidocaine group
Drug: Placebo — In the placebo group, the same volume of normal saline will be administered during anesthesia. The postoperative PCIA device will contain sufentanil 2 μg/kg, granisetron 12 mg diluted to 200 mL in 0.9% normal saline solution with a total volume of 200 mL.
  Other Names: placebo group
  Arms: Placebo group

SUMMARY:
Patients who meet the enrollment criteria will be randomized 1:1 to the lidocaine group or placebo group.

DETAILED DESCRIPTION:
Patients who meet the enrollment criteria will be randomized 1:1 to the lidocaine group or placebo group. In the lidocaine groups, lidocaine 1.5mg/kg/h was continuously infused (using ideal body weight) during the whole procedure, postoperative analgesia pump with lidocaine (lidocaine 50mg/kg, sufentanil 2ug/kg, glassetron 12mg), diluted to 200ml with saline until 72h after surgery. Blood samples will be collected from some patients in the lidocaine group for the measurement of lidocaine plasma concentration.In the placebo group, the same volume of normal saline will be administered during anesthesia. The postoperative PCIA device will contain sufentanil 2 μg/kg, granisetron 12 mg diluted to 200 mL in 0.9% normal saline solution with a total volume of 200 mL.

ELIGIBILITY:
Inclusion Criteria:

1. Participants were at least 60 years old;
2. American Society of Anesthesiologists (ASA) physical status I to III;
3. Body-mass index of 18-30 kg/m2;
4. Scheduled for elective colorectal surgery.

Exclusion Criteria:

1. Metastases occurring in other distant organs;
2. Severe hepatic insufficiency (aspartate aminotransferase or alanine transaminase or bilirubin >2.5 times the upper limit of normal);
3. Renal impairment (creatinine clearance <60 mL/min);
4. Cardiac rhythm disorders or systolic heart failure (second-and third-degree heart block, ejection fraction <50%);
5. Allergies to any of the trial drugs; chronic opioid use;
6. Inability to comprehend numeric rating scale.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Pain scores of movement-evoked pain at postoperative 24 hours | up to 24 hours postoperatively
  The pain is evaluated using numerical rating scale（NRS). NRS scores range from 0 to 10 points, with 0 points representing no pain, and 10 points representing the strongest pain.

SECONDARY OUTCOMES:
Pain scores of movement-evoked pain at postoperative 48 and 72 hours | From the date of the end of surgery until the date of 72 hours postoperatively
  The pain is evaluated using numerical rating scale（NRS). NRS scores range from 0 to 10 points, with 0 points representing no pain, and 10 points representing the strongest pain.
Pain scores of pain at rest at 24, 48 and 72 hours postoperatively | From the date of the end of surgery until the date of 72 hours postoperatively
  The pain is evaluated using numerical rating scale（NRS). NRS scores range from 0 to 10 points, with 0 points representing no pain, and 10 points representing the strongest pain.
The incidence of moderate-to-severe movement-evoked pain at 24, 48 and 72 hours postoperatively | From the date of the end of surgery until the date of 72 hours postoperatively
  The pain is evaluated using numerical rating scale（NRS). NRS scores range from 0 to 10 points, with 0 points representing no pain, 1-3 points representing mild pain, 4-6 points representing moderate pain, 7-9 points representing severe pain and 10 points representing the strongest pain.
The incidence of moderate-to-severe pain at rest at 24, 48, and 72 hours postoperatively | From the date of the end of surgery until the date of 72 hours postoperatively
  The pain is evaluated using numerical rating scale（NRS). NRS scores range from 0 to 10 points, with 0 points representing no pain, 1-3 points representing mild pain, 4-6 points representing moderate pain, 7-9 points representing severe pain and 10 points representing the strongest pain.
The cumulative morphine consumption at 24, 48, and 72 hours postoperatively | From the date of the end of surgery until the date of 72 hours postoperatively
  postoperative opioid use is reported as morphine milligram equivalents, calculated using the Practical Pain Management calculator
Time of Bowel function recovery | At 3 days after surgery
  defined as the time to first defecation or time to first flatusdefined as the time to first defecation or time to first flatus defined as the time to first defecation or time to first flatus
The incidence of postoperative nausea and vomiting during the first 72 hours postoperatively (any nausea or vomiting); | From the date of the end of surgery until the date of 72 hours postoperatively
  we considered it PONV if patients felt any nausea or had any vomiting
The incidence of a composite of postoperative pulmonary complications during hospitalisation | during the period from the end of surgery to discharge, an average of 7 days
  defined as positive if any component developed before discharge after surgery;
Length of hospital stay | during the period from the end of surgery to discharge, an average of 7 days
  Length of hospital stay
Quality of Recovery Scale Score at 24, 48, and 72 hours after surgery | From the date of the end of surgery until the date of 72 hours postoperatively
  The global QoR-15 score ranges from 0 to 150 and is categorized as five quality of recovery dimensions, including physical comfort (5 items), emotional state (4 items), psychological support (2 items), physical independence (2 items), and pain (2 items). Each piece is graded using an 11-point Likert scale. The QoR is classified according to the QoR-15 score as excellent (QoR-15 > 135), good (122 ≤ QoR-15 ≤ 135), moderate (90 ≤ QoR-15 ≤ 121) and poor (QoR-15 < 90).
Incidence of lidocaine toxicity | From the time of anesthesia induction until the date of 72 hours postoperatively
  such as new onset electrocardiogram (ECG) irregularities, drowsiness, light-headedness, metallic taste, peri-oral numbness, and tinnitus
plasma lidocaine concentration | From the time of anesthesia induction until the date of 24hours postoperatively
  Blood samples will be collected from some patients in the lidocaine group measurement of lidocaine plasma concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Weiming Li, PhD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No